CLINICAL TRIAL: NCT00454220
Title: Study to Evaluate the Dose, Safety and Effectiveness of Modified-Release Recombinant Human Thyroid Stimulating Hormone (MRrhTSH) When Used in Conjunction With Radioiodine for the Treatment of Multinodular Goiter.
Brief Title: Study to Determine the Dose, the Safety and Effectiveness of a New Drug, Modified Release rhTSH, in Patients With Multinodular Goiter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRTSH01505
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Multinodular Goiter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- 0.01 mg MRrhTSH + 131-I arm (Experimental)
  Interventions: Drug: MRrhTSH
- 0.03 mg MRrhTSH + 131-I arm (Experimental)
  Interventions: Drug: MRrhTSH

INTERVENTIONS:
Other: Placebo — 33 patients to placebo + 131-I arm
  Arms: Placebo
Drug: MRrhTSH — 33 patients to 0.01 mg MRrhTSH + 131-I arm
  Arms: 0.01 mg MRrhTSH + 131-I arm
Drug: MRrhTSH — 33 patients to 0.03 mg MRrhTSH + 131-I arm
  Arms: 0.03 mg MRrhTSH + 131-I arm

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of 2 different doses of modified-release recombinant human thyroid stimulating hormone (MRrhTSH) when administered with radioiodine in patients with multinodular goiter, a condition that involves the enlargement of the thyroid gland. We will also evaluate the safety and effectiveness of radioiodine therapy alone in these patients. The goal of the treatment is to determine if there was a reduction in the size of the goiter and to study if goiter symptoms have improved after 6 months and after 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multinodular goiter, judged clinically and by ultrasound at Screening to be at least 40 mL, but less than or equal to 140 mL in size.
* Clinically free of thyroid cancer as determined by Fine Needle Aspiration (FNA) of all dominant and/or highly suspicious cold nodules in the goiter and cytology reports as negative for thyroid cancer. (Note: Results of FNA and cytology reports that were performed within 18 months prior to commencing Screening procedures and meet these criteria are acceptable for inclusion).
* Principal Investigator must believe that there is a minimal risk of coexistent thyroid cancer.
* Principal Investigator feels that the patient's iodine intake and/or levels will not significantly impact the results of the study (urinary iodine assay at Screening and low-iodine diet are optional and associated data will not be collected for study purposes).
* Baseline serum level of free thyroxine index (FTI) within the normal range, as determined by central lab.
* Baseline serum level of thyroid stimulating hormone (TSH) ranges from undetectable to the upper limit of the normal range, as determined by central lab.
* Females of child-bearing potential must be on a stable hormonal contraceptive regimen (i.e., > 6 months continuous use) and/or use a double barrier method (i.e., condom and foam) through Visit 8 (i.e. the end of the Core Study).
* Through Visit 8 (6 months) of a male patient's participation in the study, it is recommended that his sexual partner(s), who are females of child-bearing potential, use the above described methods of contraception.
* Negative pregnancy tests for all women of child-bearing potential prior to participating in the study. Women aged 50 years and above and considered postmenopausal (defined as > 2 years since last menstrual period) will not need to have a pregnancy test.
* Routine blood laboratory values within normal range at Screening, as determined by central lab. Abnormal values considered to be not clinically significant by the Principal Investigator are acceptable for inclusion.
* Electrocardiogram (ECG) (12 lead, 2 minute rhythm strip) within normal limits at Screening as determined by a designated study cardiologist or appropriately qualified physician at each site. Evidence of an old myocardial infarction (MI) will exclude the patient. Patients who have ECG findings of occasional premature atrial beats, abnormal PR intervals not associated with supra ventricular tachycardia (SVT) or heart block, right bundle branch block, and heart rates ≤ 100 beats per minute (BPM) and ≥ 50 BPM may be included in this study.
* Committed to follow all protocol-required study procedures as evidenced by providing written informed consent within 21 days prior to Screening Period 2.

Exclusion Criteria:

* History of thyroid cancer.
* Previous partial or near total thyroidectomy.
* Clinical history, signs or symptoms that make thyroid cancer a higher than usual probability, such as positive immediate family history of thyroid cancer, history of head or neck irradiation, a stone-hard nodule or suspicious growth of a nodule in recent months, palpable cervical lymph nodes or nodes that on ultrasound have features suspicious for metastases (unless ruled out by biopsy or FNA).
* During the 45 days before administration of MRrhTSH or placebo (i.e., Screening Periods 1 and 2), use of propylthiouracil, methimazole or thyroxine, vitamins or supplements containing kelp or iodine (taking a multivitamin that does not contain iodine or kelp is acceptable), medications that significantly affect iodine handling such as high dose corticosteroids, high dose diuretics, or lithium (low or moderate dose diuretic use is acceptable).
* Patient has currently or within the past 60 days used retinoic acid.
* Serum calcitonin above the upper limit of normal at Screening, as determined by central lab.
* Use of amiodarone within the prior 2 years.
* Received iodine-containing contrast agent within the past 3 months.
* Inability to complete all required visits.
* Patients with conditions in which use of beta-blockers are medically contraindicated, such as recently active asthma or clinically significant chronic obstructive pulmonary disease.
* Currently or within the past 5 years have a history of malignancy, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Prior MI, even if remote; stroke within 6 months; atrial fibrillation or clinically significant arrhythmia within 6 months (patient may have mild hypertension or chronic cardiac illnesses that are well controlled on a medication regimen: blood pressure (BP) less than 140/90 mmHg after resting 5 minutes).
* A concurrent major medical disorder (e.g., documented significant cardiac disease, debilitating cardiopulmonary disease, advanced renal failure, advanced liver disease, advanced pulmonary disease, or advanced cerebral vascular disorder) that may have an impact on the capability of the patient to adequately comply with the requirements of this study.
* Women who are pregnant or lactating.
* A recent history of alcoholism, drug abuse or other disorder that might affect compliance with the protocol.
* Received investigational study medication within 30 days prior to signing informed consent and/or intends to participate in another clinical study involving the use of an investigational drug over the course of study participation.
* Patients on anticoagulants except for aspirin.
* Patients known at the time of Screening due to past testing to be human immunodeficiency virus (HIV) antibody positive or hepatitis B antigen positive (no screening for HIV or hepatitis B should be done in the study).
* Hyperthyroid symptom scale (HSS) ≥ 20.
* Patients who have received 131I in the past, and have had a lifetime exposure believed to be >10 mCi (0.37GBq) of 131I.
* History of allergy to Thyrogen.
* Sodium carboxymethylcellulose (NaCMC) allergy (including prior history of anaphylaxis following topical lidocaine, barium sulfate ingestion, or intra-articular or parenteral corticosteroid).
* Smallest cross-sectional area of the trachea (SCAT) discovered on CT to be < 60 mm2

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months in goiter size by computer tomography (CT) scan. | Duration of core study
Extension Phase: Change in goiter size by CT scan at 36 months versus baseline, Months 6, 12 and 24 | Duration of extension phase

SECONDARY OUTCOMES:
Change in goiter size from baseline to 6 months in smallest cross sectional area of the trachea (SCAT). | Duration of core study
The percentage of patients in each group who attained a goiter volume shrinkage at 6 months of 28% or greater. | Core Study
Extension Phase: Change in goiter size from baseline to 6, 12, 24 and 36 months by SCAT and neck ultrasound. | Duration of extension phase
Thyroid Quality of Life Questionnaire | Core Study and Extension Phase
Thyroid Stimulating Hormone (TSH), free thyroxine (FT4), total thyroxine (TT4), FT1, free triiodothyronine (FT3), total T3 (TT3). | Core Study and Extension Phase
Physical Exams, Vitals, Adverse Events, Respiratory symptoms | Core Study and Extension Phase
Routine labs, serial thyroid function tests, antibodies to MRrhTSH, antibodies against the thyroid stimulating hormone receptor, and physical exam. | Core study and extension phase
Tracheal diameter measurements determined by ultrasound at Visit 3 compared to baseline measurement. | core study - Visit 3
Electrocardiogram (ECG) | Duration of core study
Treatment-emergent hyperthyroidism (Hyperthyroid Symptom Scale (HSS) score ≥ 20). | Core study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (11):
- Boston, Massachusetts, United States
- Brazil (2):
  - Curitiba
  - Rio de Janeiro
- Canada (2):
  - London, Ontario
  - Toronto
- Odense, Denmark
- Lille, France
- Würzburg, Germany
- Italy (2):
  - Pisa
  - Siena
- Netherlands, Netherlands

REFERENCES:
- [Result] Fast S, Hegedus L, Pacini F, Pinchera A, Leung AM, Vaisman M, Reiners C, Wemeau JL, Huysmans DA, Harper W, Rachinsky I, de Souza HN, Castagna MG, Antonangeli L, Braverman LE, Corbo R, Duren C, Proust-Lemoine E, Marriott C, Driedger A, Grupe P, Watt T, Magner J, Purvis A, Graf H. Long-term efficacy of modified-release recombinant human thyrotropin augmented radioiodine therapy for benign multinodular goiter: results from a multicenter, international, randomized, placebo-controlled, dose-selection study. Thyroid. 2014 Apr;24(4):727-35. doi: 10.1089/thy.2013.0370. Epub 2014 Mar 4. PMID 24341527
- [Derived] Huo Y, Xie J, Chen S, Wang H, Ma C. Recombinant human thyrotropin (rhTSH)-aided radioiodine treatment for non-toxic multinodular goitre. Cochrane Database Syst Rev. 2021 Dec 28;12(12):CD010622. doi: 10.1002/14651858.CD010622.pub2. PMID 34961921